CLINICAL TRIAL: NCT06756672
Title: Hypotension Prediction Index for Prevention of Hypotension and Postoperative Complications During Laparoscopic Surgery for Colorectal Cancer: A Multi-Center Randomized Trial
Brief Title: HPI in Laparoscopic Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202408037DINB
Record Dates: First submitted 2024-12-15; First posted 2025-01-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-11

CONDITIONS: the Duration and Severity of Intraoperative Hypotension
Keywords: Hypotension Prediction Index; intraoperative hypotension; laparoscopic colorectal surgery

STUDY DESIGN:
Intervention Model Description: patients undergoing hypotension prediction index guidance
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not know which group they are in, nor will the outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI guidance (Experimental): patients with HPI guidance
  Interventions: Device: HPI guidance
- patients in the control group (Active Comparator): patients without HPI guidance
  Interventions: Device: No HPI guidance

INTERVENTIONS:
Device: HPI guidance — patients with HPI guidance
  Arms: HPI guidance
Device: No HPI guidance — patients without HPI guidance
  Arms: patients in the control group

SUMMARY:
Using the Hypotension Prediction Index in patients undergoing laparoscopic colorectal surgery, including data from National Taiwan University Hospital and Taipei Veterans General Hospital

DETAILED DESCRIPTION:
Intraoperative hypotension is a common occurrence during laparoscopic colorectal cancer resection, often attributable to factors such as general anesthesia, the growing population of elderly patients, and the use of pneumoperitoneum during surgery. This condition, defined as a mean arterial pressure (MAP) below 65 mmHg, is linked to major organ complications within 30 days postoperatively. Introduced in 2019, the Hypotension Prediction Index (HPI) is an algorithm designed to predict the onset of intraoperative hypotension. Previous studies have used the time-weighted average MAP below 65 mmHg as a primary endpoint, calculated as the area under the MAP curve <65 mmHg (mmHg × hours) divided by the duration of surgery (hours), with a value ≥0 indicating severity. Higher values reflect more severe hypotension. However, research on the application of HPI in laparoscopic colorectal cancer resection remains limited. This study aims to determine whether the use of HPI can reduce the severity of intraoperative hypotension in patients undergoing laparoscopic colorectal cancer resection and whether it can decrease the incidence of major postoperative organ complications. A total of 120 patients, aged 20-80 years and undergoing elective laparoscopic colorectal cancer resection, will be randomly assigned to two groups: an intervention group guided by HPI and a control group without HPI guidance. In the intervention group, an alert will be triggered when the HPI exceeds 85, indicating a potential MAP drop below 65 mmHg, whereas the control group will initiate hypotension treatment only when MAP falls below 65 mmHg. Both groups will adhere to the same intraoperative hypotension management protocols, including fluid resuscitation, vasopressor administration, and observation. The primary treatment outcome will be the time-weighted average MAP <65 mmHg, and major postoperative organ complications will be monitored for 30 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective laparoscopic colorectal surgery

Exclusion Criteria:

* Severe heart or lung diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
time weighted average mean arterial pressure (TWA MAP) <65 mmHg (unit: mmHg) | during the whole surgery
  the severity and duration of hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital and Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to ethical issue